CLINICAL TRIAL: NCT00285532
Title: Identifying Residential Hazards Using Home Test Kits
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 11261-CP-002
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Poisoning, Lead
Keywords: Blood Lead; Pesticides; Community-based; Sampling Kits
MeSH Terms: conditions — Lead Poisoning

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Home test kit

SUMMARY:
The purpose of this project is to help families and communities identify and reduce health risks from lead, pesticides and, ultimately, other environmental hazards. We have partnered with the Better Housing League and Baby's Milk Fund in Cincinnati and nationally with the Alliance to End Childhood Lead Poisoning and the National Center for Lead Safe Housing. The first specific aim of this project is to evaluate a sampling kit for families to assess levels of lead and pesticides in their home environment. This aim will strengthen right-to-know laws by providing families with tools to assess environmental contamination in their own homes. The second aim is to increase community awareness of the role of environmental agents in developmental disorders, hearing loss and school problems.

DETAILED DESCRIPTION:
A cross-sectional random, stratified study design will be used for this project. All children who are younger than 5 years of age and have a venipuncture blood sample taken at the babies Milk Fund Clinic will be eligible for this study. After checking the lists for errors and duplications, we will randomly permute the sampling frame, stratifying on children's blood lead concentration. Stratification will be used to enroll about 33% of the sample with blood lead concentrations below 5 mg/dl, 33% between 5 to 10 mg/dl, and 33% of 10 mg/dl or higher. Stratifying the sample will improve our chances of testing the predictive validity of home sampling kits to identify children who have blood lead concentration > 10 mg/dl collected by families. In addition this study will:

1. Develop a pesticide wipe sampling kit to accompany our lead-sampling kit.
2. Evaluate the predictive validity of home sampling kits for lead-contaminated floor dust to identify children who have blood lead levels of 10 mg/dl or higher by community participants compared with repeat samples taken by trained, community workers.
3. Evaluate the reliability of home sampling kits for pesticides in dust collected by community participants compared with trained, community workers.
4. Disseminate data on the reliability of home sampling tests and provide tools for families to collect environmental samples for large, population-based studies.
5. Develop a Healthy Homes Resource Center at the Better Housing League to disseminate information to the community about residential hazards.

ELIGIBILITY:
Inclusion Criteria:

Venous blood lead In residence 3 months Child less than 5 years of age Sampler greater than 18 years of age

Exclusion Criteria:

Cannot read or understand English Physically unable to conduct field sampling Outside of theGreater Cincinnati area

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children <5 years receiving care via Babies Milk Fund Clinics
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2001-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Lead and Pesticide Levels | One time home visit 3-5 days after distribution of kits

CONTACTS AND LOCATIONS:
Overall Officials: Sandy M Roda, BS, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States